CLINICAL TRIAL: NCT01231672
Title: Evaluation and Prospective Validation of Clini-biological Parameters Including Initial Hemostasis, Which Improve the Prediction of Death at 1 Month Among Patients Entering Intensive Care Units for Septic Shock
Brief Title: Prospective Validation of Clini-biological Parameters Including Initial Hemostasis, Which Improve the Prediction of Death at 1 Month Among Patients With Septic Shock
Acronym: SEPSICOAG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2008/GL-03; 2008-A01214-51 (Other: ANSM)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Shock, Septic
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Septic shock patients
  Interventions: Biological: Routine biological analyses

INTERVENTIONS:
Biological: Routine biological analyses — Bilirubinemia (total and conjugated), hematology, hemogram, SOFA score

SUMMARY:
A prognostic score was proposed by the investigative team to predict death at 1 month. This score is based on certain biological markers, scored under emergency conditions in the first 24 hours of routine clinical practice management for septic shock.

The main objective of this multicenter study is to validate the performance of the score in terms of area under the ROC curve and negative predictive value.

DETAILED DESCRIPTION:
There are two secondary objectives:

* Validate a prognostic score for death at the end of the first week from initial data.
* Validate a predictive score of disseminated intravascular coagulation (DIC) in patients with septic shock by comparing with the Gold Standard of the International Society on Thrombosis and Haemostasis (overt-DIC in the first 5 days after inclusion).

As for the main objective, these scores are based on biological markers scored under emergency situations within the first 24 hours of routine clinical practice management for septic shock.

The objectives and endpoints stated correspond to the protocol directly submitted to ethics authorities prior to the first inclusion and can be verified by contacting the Committee for the Protection of Persons Sud Mediterranée III (mail: CPP SUD-MEDITERRANEE III, UFR MEDECINE 186, chemin du Carreau de Lanes CS 83021, 30908 NIMES Cedex 2 FRANCE. Study reference: 2008.11.04 bis) For more information: carey.suehs@chu-nimes.fr

ELIGIBILITY:
Inclusion Criteria:

* patient (or representative) received the information notice
* patient has hemodynamic insufficiency of non-traumatic or cardiogenic origin associated with severe sepsis (treated with Noradrenalin) and organ dysfunction, hypoperfusion or hypotension
* body temperature > 38.3°C or < 36°C
* heart rate > 90 bpm
* Tachypnea > 20 C/min or PaCO2 < 32 mmHg or mechanical ventilation
* leukocytes > 12000 µL-1 ou < 4000 µL-1 ou > 10% immature forms
* oliguria < 0.5 ml/kg/h for at least 2 hours
* abrupt alteration (24 h) of conscienceness
* thrombocytopenia < 100 000 G/L or disseminated intravascular coagulation
* mottled skin and / or capillary refill time> 3 sec
* PaO2/FiO2 < 300 mmHg ou < 40KPas
* Lactatemia > 2mMol/l
* septic shock: Systolic Blood Pressure (SBP) > 90 mmHg or need for vasopressors to maintain SBP> 90 mmHg despite a prior filling (20-30 ml / kg of macromolecules or 40 to 60 ml / kg of normal saline (or decrease in SBP> 40% in the hypertensive)

Exclusion Criteria:

* patient is dying or limitation or cessation of active treatment
* patient is already included in another trial
* patient or family refusal
* patient not affiliated with a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe septic shock patients entering intensive care units in the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2009-04; Primary Completion 2013-10-30 (Actual); Study Completion 2013-10-30 (Actual)

PRIMARY OUTCOMES:
AUC of the studied prognostic score | 24 hours (studied score parameters); 1 month (mortality)
  The biological parameters measured at the time of admission to the intensive care unit and that make up the prognostic score for death at 1 month will be collected. The event "death within 1 month" will be analyzed. For patients discharged from service before the end of the first month, the clinician will still be informed concerning possible death.
  The studied biological parameters correspond to routine coagulation and hematological parameters for patients in septic shock, according to SFAR (Société Française d'Anesthésie et de Réanimation) recommendations and the SRLF (Société de Réanimation de Langue Française) Consensus (2002).
Negative predictive value of the studied prognostic score | 24 hours (studied score parameters); 1 month (mortality)
  The biological parameters measured at the time of admission to the intensive care unit and that make up the prognostic score for death at 1 month will be collected. The event "death within 1 month" will be analyzed. For patients discharged from service before the end of the first month, the clinician will still be informed concerning possible death.
  The studied biological parameters correspond to routine coagulation and hematological parameters for patients in septic shock, according to SFAR (Société Française d'Anesthésie et de Réanimation) recommendations and the SRLF (Société de Réanimation de Langue Française) Consensus (2002).

SECONDARY OUTCOMES:
AUC of the studied prognostic score | 24 hours (studied score parameters); 1 week (mortality)
  Biological parameters at the time of intensive care unit admission and making up the prognostic score for death at 1 week will be collected. The event "death within 1 week" will be analyzed. For patients discharged from the department before the end of the first week, the clinician will still be informed of possible death. For the prognostic score at 1 week, a single biological parameter is used: fibrinogen. Age and SAPSII are also included in the score.
Negative predictive value of the studied prognostic score | 24 hours (studied score parameters); 1 week (mortality)
  Biological parameters at the time of intensive care unit admission and making up the prognostic score for death at 1 week will be collected. The event "death within 1 week" will be analyzed. For patients discharged from the department before the end of the first week, the clinician will still be informed of possible death. For the prognostic score at 1 week, a single biological parameter is used: fibrinogen. Age and SAPSII are also included in the score.
AUC of the studied prognostic score | 24 hours (studied score parameters); 5 days (DIC)
  Our secondary objective is to validate a clinicobiological score, including hemostasis parameters (clotting factors and coagulation activation) and a clinical score (SOFA) for predicting the occurrence of DIC in the first 5 days after inclusion.
  The DIC score will be calculated according to ISTH (International Society on Thrombosis and Haemostasis) recommandations (Taylor et al, 2001).
Negative predictive value for the studied prognostic score | 24 hours (studied score parameters); 5 days (DIC)
  Our secondary objective is to validate a clinicobiological score, including hemostasis parameters (clotting factors and coagulation activation) and a clinical score (SOFA) for predicting the occurrence of DIC in the first 5 days after inclusion.
  The DIC score will be calculated according to ISTH (International Society on Thrombosis and Haemostasis) recommandations (Taylor et al, 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Lavigne-Lissalde, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (7):
- France (7):
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - APHM - Hôpital de la Conception, Marseille
  - AP-HM Hôpital Nord, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CHU de Nice, Nice
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - CHU de Saint Etienne, Saint-Etienne

REFERENCES:
- [Result] Gris JC, Faillie JL, Cochery-Nouvellon E, Lissalde-Lavigne G, Lefrant JY. ISTH overt disseminated intravascular coagulation score in patients with septic shock: automated immunoturbidimetric soluble fibrin assay vs. D-dimer assay. J Thromb Haemost. 2011 Jun;9(6):1252-5. doi: 10.1111/j.1538-7836.2011.04270.x. No abstract available. PMID 21645228